CLINICAL TRIAL: NCT06498219
Title: Optimization of the Skin Test Procedure With Iodinated Contrast Products for Certain Patients Suspected of Immediate Hypersensitivity
Acronym: OPT-TC-PCI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9025
Record Dates: First submitted 2024-07-04; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Contrast Sensitivity
Keywords: Contrast Sensitivity; Iodinated contrast products; Allergic immunological mechanisms; Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypersensitivity to iodinated contrast products (ICP) affects 1 to 3% of injected patients. These reactions require an allergological assessment with skin tests in order to distinguish allergic immunological mechanisms from other non-specific mechanisms. Current recommendations recommend carrying out prick tests followed by intradermal reactions up to a 10th dilution. However, undiluted IDRs are carried out by several teams under certain conditions, without this having been validated. Experience tends to show that these IDRs are relevant in certain patients to make the diagnosis without risk.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Subject treated in the allergology department in the period from June 1, 2020 to July 3, 2023 for suspected allergic hypersensitivity to ICPs and having had at least one undiluted intradermal reaction to one or more ICPs.
* Absence of written opposition in the medical file of the subject (and/or their legal representative if applicable) to the reuse of their data for scientific research purposes.

Exclusion Criteria:

* Presence of opposition from the subject (and/or their legal representative if applicable) to the reuse of their data for scientific research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old) treated in the allergology department in the period from June 1, 2020 to July 3, 2023 for suspected allergic hypersensitivity to ICPs and having had at least one undiluted intradermal reaction to one or more ICPs.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of the relevance of performing pure intradermal reactions to iodinated contrast products (ICP) after obtaining a pure negative prick test. | Files analyzed retrospectively cover the period from June 1, 2020 to July 3, 2023.
  This retrospective study concerns patients treated at the Strasbourg University Hospital in the period from June 1, 2020 to July 3, 2023 for suspected allergic hypersensitivity to (ICP) and having had at least one undiluted intradermal reaction to one or more (ICP) .

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pneumologie - CHU de Strasbourg - France, Strasbourg, France